CLINICAL TRIAL: NCT06844292
Title: Evaluation of Microinvasive Glaucoma Surgery: MINIject® Versus Hydrus® Microstent in Combination With Cataract Surgery
Acronym: MINHY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1242/2024
Record Dates: First submitted 2025-02-06; First posted 2025-02-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma; Cataract
Keywords: Glaucoma; Open-angle Glaucoma; Cataract; Minimally Invasive Glaucoma Surgery (MIGS); Intraocular Pressure (IOP) Reduction
MeSH Terms: conditions — Glaucoma; Cataract; Glaucoma, Open-Angle | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Device: Phacoemulsification combined with minimally invasive glaucoma surgery (MIGS), either Hydrus Microstent or MINIject. The patients will be randomized (1:1) to each treatment/intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MINIject (Active Comparator): MINIject with Cataract Surgery
  Interventions: Device: MINIject with Cataract Surgery
- Hydrus Microstent (Active Comparator): Hydrus Microstent with Cataract Surgery
  Interventions: Device: Hydrus Microstent with Cataract Surgery

INTERVENTIONS:
Device: MINIject with Cataract Surgery — Patients will be randomized to receive either a MINIject implant or a Hydrus Microstunt in conjunction with cataract surgery. If randomized to MINIject, the device will be implanted into the supraciliary space with a minimally invasive ab interno approach. It is designed to be implanted with its head in the anterior chamber and its body in the supraciliary space, leading to improved natural uveoscleral outflow by directing aqueous humor from the anterior chamber to the sub-scleral space. Cataract surgery will be performed with phacoemulsification.
  Arms: MINIject
Device: Hydrus Microstent with Cataract Surgery — Patients will be randomized to receive either a Hydrus Microstunt or a MINIject implant in conjunction with cataract surgery. If randomized to Hydrus Microstent, the device will be implanted into Schlemm's canal through the trabecular meshwork in order to dilate and restore the natural aqueous outflow pathway through Schlemm's canal, leading to a reduction of intraocular pressure.
  Cataract surgery will be performed with phacoemulsification.
  Arms: Hydrus Microstent

SUMMARY:
The study aims to investigate postoperative outcomes after two different MIGS implants (MINIject or Hydrus) in combination with cataract surgery for patients with glaucoma.

DETAILED DESCRIPTION:
The study aims to investigate postoperative outcomes in terms of intraocular pressure as well as safety measures after two different MIGS implants (MINIject® or Hydrus®) in conjunction with cataract surgery (CS) for patients with chronic glaucoma. The patients will be followed up for 5 years after the date of their implantation. Standard ophthalmologic assessments including measurement of intraocular pressure, fundus examination and ocular imaging with OCT (Optical Coherence Tomography). Assessment of life quality as well as adverse events will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma in which surgery is indicated to reach target intraocular pressure as well as lens opacities where CS is indicated
* Clinically eligible for both surgeries
* Subjects not anticipated to require any further surgery in the next 12 months
* Patients' age > 18 years

Exclusion Criteria:

* Patients who do not want to make follow-ups at the department
* Angle closure, uveitic, neovascular, congenital glaucoma, iridocorneal endothelial syndrome, Axenfeld-Rieger syndrome
* Prior filtering glaucoma surgery, suprachoroidal stent, retinal surgery, corneal graft surgery or cyclophotocoagulation
* Allergy to any drugs or substances required for the protocol
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-03-03 (Estimated); Study Completion 2031-03-03 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure After Surgery | Baseline visit to 1 year
  Mean IOP in mmHg one year after glaucoma surgery

SECONDARY OUTCOMES:
Intraocular Pressure at Other Follow-Up Time Points | Baseline visit to 5 years
  IOP at other follow-up visits such as week 1, month 1/3/6 and year 2/3/4/5 after surgery.
Anti-Hypertensive Medications Required | Baseline visit and week 1, month 1/3/6 and year 1/2/3/4/5
  Number and type of anti-hypertensive medications used at specific study visit
Best Corrected Visual Acuity | Baseline visit and week 1, month 1/3/6 and year 1/2/3/4/5
  Best Corrected Visual Acuity will be measured with Snellen charts and will be transformed to logMAR.
Complete Success | Baseline visit and visit at month 3/6 and year 1/2/3/4/5
  Complete success is defined as either unmedicated IOP ≤21 mmHg, ≤18 mmHg, ≤15 and ≤12 mmHg and >5 mmHg
Qualified Success | Baseline visit and visit at month 3/6 and year 1/2/3/4/5
  Qualified success is defined as either medicated IOP ≤21 mmHg, ≤18 mmHg, ≤15 and ≤12 mmHg and >5 mmHg
Endothelial Cell Density | Baseline visit and visit at year 1/2/3/4/5
  Endothelial cell density will be measured with a specular microscope.
Assessment of Life Quality - Glaucoma Quality of Life-15 Questionnaire | Baseline visit and visit at month 6 and year 1/2/3/4/5
  A modified Glaucoma Quality of Life-15 (GQL-15) Questionnaire will be used to determine and document quality of life. The GQL-15 questionnaire is a 15-item survey designed to assess the impact of glaucoma on a patient's daily life and well-being. It evaluates how symptoms like vision impairment, discomfort, and treatment affect daily activities. The scores range from 0 (Minimum) to 60 (Maximum), with higher scores indicating a greater negative impact on quality of life, while lower scores suggest less impairment.
  0-15: Minimal impact on quality of life 16-30: Mild impact on quality of life 31-45: Moderate impact on quality of life 46-60: Severe impact on quality of life
Assessment of Life Quality - Ocular Surface Disease Index | Baseline visit and visit at month 6 and year 1/2/3/4/5
  The Ocular Surface Disease Index (OSDI) will be used to determine and document quality of life. The OSDI is a 12-item questionnaire used to assess the severity of dry eye symptoms and their impact on daily life. The total score ranges from 0 (Minimum) to 100 (Maximum), with higher scores indicating more severe symptoms.
  0-12: Minimal or no dry eye symptoms 13-22: Mild symptoms 23-32: Moderate symptoms 33-100: Severe symptoms
Rate of Additional Ocular Surgery Post-Implantation | 5 years
  Rate of additional ocular surgery post-implantation will be collected at every study visit.
Rate of Complications or Incidents | 5 years
  Complications associated with both surgical procedures will be assessed.
Data From Optical Biometry - Axial Length | Baseline visit and year 1 visit
  Axial Length of the eyeball from optical biometry will be measured.
Data From Optical Biometry - Anterior Chamber Depth | Baseline visit and year 1 visit
  Anterior chamber depth from optical biometry will be measured.
Data From Optical Biometry - Corneal Surface Parameters | Baseline visit and year 1 visit
  Corneal surface parameters (K-values) from optical biometry will be measured.
Standard Automated Perimetry | Baseline visit and visit at month 6 and year 1/2/3/4/5
  Standard automated perimetry will be examined, the mean defect will be given in dB.
Optical Coherence Tomography - RNFL Thickness | Baseline visit and visit at month 1/3/6 and year 1/2/3/4/5
  RNFL (retinal nerve fiber layer) thickness will be measured via OCT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Ewald Lindner, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No
not necessary